CLINICAL TRIAL: NCT03748745
Title: A Single-center, Open-label, Steady-state Drug-drug Interaction Study of SH229 Tablets and Daclatasvir Dihydrochloride Tablets in Healthy Subjects
Brief Title: A Drug-drug Interaction Study of SH229 Tablets and Daclatasvir Dihydrochloride Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Sanhome Pharmaceutical, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SHC005-I-04
Record Dates: First submitted 2018-11-02; First posted 2018-11-21 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Drug Interactions
Keywords: HCV; SH229
MeSH Terms: interventions — daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): SH229 (600 mg) once daily, Daclatasvir dihydrochloride (60 mg) once daily.
  Interventions: Drug: SH229; Drug: Daclatasvir dihydrochloride
- Cohort B (Experimental): SH229 (600 mg) once daily, Daclatasvir dihydrochloride (60 mg) once daily.
  Interventions: Drug: SH229; Drug: Daclatasvir dihydrochloride

INTERVENTIONS:
Drug: SH229 — tablet, oral, 600 mg once daily for day 1 to day 14
  Arms: Cohort A
Drug: SH229 — tablet, oral, 600 mg once daily for day 8 to day 14
  Arms: Cohort B
Drug: Daclatasvir dihydrochloride — tablet, oral, 60 mg once daily for day 8 to day 14
  Arms: Cohort A
Drug: Daclatasvir dihydrochloride — tablet, oral, 60 mg once daily for day 1 to day 14
  Arms: Cohort B

SUMMARY:
The purpose of this study is to evaluate the drug-drug interaction of SH229 tablets and Daclatasvir dihydrochloride tablets. The study also evaluates the pharmacokinetics and tolerability of co-administration of SH229 tablets and Daclatasvir dihydrochloride tablets in healthy subjects. This study provides evidence for the designing of following clinical trial protocols.

DETAILED DESCRIPTION:
A total of 28 evaluable healthy subjects will be enrolled in this study. The dose of SH229 is 600 mg. The dose of Daclatasvir dihydrochloride is 60 mg.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form before the study and fully understand the study content, process and possible adverse reactions;
2. Be able to complete the study as required by the protocol;
3. Subjects (including their partners) who are willing to voluntarily take effective contraceptive measures from screening to 6 months after the last dose. See the appendix for specific contraceptive measures;
4. Male subjects aged 18-45 (including 18 and 45 years old);
5. Male subjects who weigh no less than 50 kg and have a body mass index between 18 and 28 kg / m2 (including the threshold). Body mass index (BMI) = weight (kg) / height2 (m2);
6. Physical examination and vital signs normal, or the abnormal signs have no clinical significance.

Exclusion Criteria:

1. Smoke more than 5 cigarettes per day within three months prior to study;
2. Subjects who are allergic to the study drugs or prone to allergies (Multiple drug and food allergies);
3. Subjects with history of drug and/or alcohol abuse (14 units per week: 1 unit = 285 mL of beer, or 25 mL of hard liquor, or 100 mL of wine);
4. Subjects with history of blood donation or massive blood loss (> 450 mL) within three months prior to screening;
5. Subjects with dysphagia or have history of gastrointestinal disorders which affects study drug absorption;
6. Subjects with any diseases that increase the risk of bleeding, such as hemorrhoids, acute gastritis, or gastric and duodenal ulcers;
7. Use of any drugs that alter liver enzyme activity within 28 days prior to screening;
8. Use of any prescription drugs, over-the-counter drugs, vitamin products or herbal medicines within 14 days prior to screening;
9. Use of special diet (including dragon fruit, mango, grapefruit, etc.), strenuous activities or other factors that may affect the absorption, distribution, metabolism and excretion of the study drug within 2 weeks prior to screening;
10. Concomitant use of strong inhibitors or inducers of CYP3A4, P-gp or Bcrp, such as itraconazole, ketoconazole or dronedarone;
11. Subjects with major changes in diet or exercise habits recently;
12. Use of study drugs or participation in other clinical trials within three months prior to dosing;
13. Subjects who have ECG abnormalities with clinical significance;
14. Subjects who have abnormalities with clinical significant in clinical laboratory tests or other clinical findings that indicate clinically significant diseases (including but not limited to gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric or cardiovascular diseases);
15. Subjects with viral hepatitis (including hepatitis B and hepatitis C), AIDS antibody and/or antibody screening positive for Treponema pallidum;
16. Subjects with acute disease or concomitant use of drugs from screening stage to dosing;
17. Use of chocolate, food or beverages containing caffeine or xanthine within 24 hours prior to dosing;
18. Use of products containing alcohol within 24 hours prior to dosing;
19. Subjects with urine drug screening test positive, or with history of drug abuse in the past 5 years;
20. Subjects with any other reasons that investigator considers to be unsuitable for the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2018-12-25 (Actual); Study Completion 2018-12-25 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 1 month after last dose
  Cohort A and Cohort B [Safety and tolerability]

SECONDARY OUTCOMES:
Tmax, ss | Day 5, 6, 7, 8, 12, 13, 14, 15, 16, 17 after first dose
  Time of maximum observed concentration; safety and validity criteria
Cmax, ss | Day 5, 6, 7, 8, 12, 13, 14, 15, 16, 17 after first dose
  Maximum observed concentration; safety and validity criteria
Cmin, ss | Day 5, 6, 7, 8, 12, 13, 14, 15, 16, 17 after first dose
  Minimum observed concentration; safety and validity criteria
t1/2, ss | Day 5, 6, 7, 8, 12, 13, 14, 15, 16, 17 after first dose
  Elimination half-life; safety and validity criteria
AUC0-24, ss | Day 5, 6, 7, 8, 12, 13, 14, 15, 16, 17 after first dose
  Area under the concentration-time curve (AUC) from time 0 to 24 hours; safety and validity criteria
AUC0-72, ss | Day 5, 6, 7, 8, 12, 13, 14, 15, 16, 17 after first dose
  Area under the concentration-time curve (AUC) from time 0 to 72 hours; safety and validity criteria
AUC0-∞, ss | Day 5, 6, 7, 8, 12, 13, 14, 15, 16, 17 after first dose
  Area under the concentration-time curve (AUC) from time 0 to infinity; safety and validity criteria
CL/F ss | Day 5, 6, 7, 8, 12, 13, 14, 15, 16, 17 after first dose
  Apparent clearance; safety and validity criteria
DF | Day 5, 6, 7, 8, 12, 13, 14, 15, 16, 17 after first dose
  Degree of fluctuation; safety and validity criteria

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, MD, Principal Investigator — Phase I Clinical Trial Unit, The First Hospital of Jilin University
Locations (1):
- Phase I Clinical Trial Unit, The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No